CLINICAL TRIAL: NCT06278506
Title: Resection or Ablative Treatment of Small Renal Tumors, a Multicenter Randomized Clinical Trial
Brief Title: Resection or Ablation of Small Kidney Tumors
Acronym: RESTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Kjellman, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4612
Record Dates: First submitted 2024-01-30; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Radiofrequency Ablation; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation (Experimental): Ablative treatment of small kidney cancer lesion, could be given with radiofrequency, microwawe or cryoablation
  Interventions: Procedure: Ablation
- Partial nephrectomy (Active Comparator): Surgical resection with open or laparoscopic technique
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Ablation — Microwave ablation, Radiofrequency ablation, Cryo ablation
  Other Names: Microwave ablation, Radiofrequency ablation, Cryo ablation
  Arms: Ablation
Procedure: Surgery — Partial or total nefrectomy
  Other Names: Partial nefrectomy, total nefrectomy
  Arms: Partial nephrectomy

SUMMARY:
Ablative treatments are believed to have a lower rate of complications, shorter hospital stays, and fewer interventions with benign PAD compared to partial nephrectomies in small kidney cancer lesions. The purpose of the study is to compare complications, the frequency of residual tumors, impact on kidney function, differences in quality of life, and health economic factors in a randomised study. We will also compare the oncological outcomes, including survival and recurrence of kidney cancer.

DETAILED DESCRIPTION:
Kidney cancer represents approximately 2-3% of all cancer cases, with about 400,000 new cases and 175,000 deaths worldwide in 2018. In Sweden, about 1,200 new cases of kidney cancer are detected each year. The most common age for diagnosis is between 60 and 80 years, and it is more prevalent in men than in women. Many cases are incidentally discovered during imaging studies for unrelated issues. There has been an increase in incidentally detected tumors in Sweden, from 43% in 2005 to 69% in 2021. Nephron-sparing surgery, i.e., partial nephrectomy, is recommended for preserving kidney function in localized tumors.

Ablative treatments are recommended for patients with significant comorbidities, multiple tumors, a single kidney, or other situations where surgery is not considered suitable. Prior to treatment, a biopsy is usually performed to confirm the diagnosis. Studies show variations in oncological outcomes based on the subgroups of kidney cancer treated with ablative techniques. Ablative techniques seem to have a lower risk of complications compared to surgery concerning perioperative complications, bleeding, and maintaining kidney function for a longer time. However, there are no randomized controlled studies comparing ablative treatment with nephrectomy for T1a tumors in the kidney.

3. Hypothesis

Ablative treatment of small kidney tumors may result in shorter hospital stays with fewer complications compared to surgical resection.

There is no difference in long-term oncological outcomes between the methods.

4. Outcome Measures

The primary purpose of the study is to compare surgical complications, findings of remaining tumors after primary treatment, and the time patients are hospitalized after each procedure. Secondary outcomes include oncological outcomes in the short and long term, as well as functional factors

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 99 years
* Patient suitable based on clinical status for both ablative treatment and surgery
* Primary kidney tumor
* Tumor size ≤ 3 cm
* Clinical stage of the tumor T1a (no macroscopic vascular or extrarenal invasion)
* Tumor location suitable for both ablative treatment and resection
* Absence of radiological signs of metastasis
* Biopsy with malignant pathological analysis (PAD)
* ISUP grade I-III"

Exclusion Criteria:

* Radiological signs of metastasis
* Synchronous kidney tumors
* ISUP grade IV or sarcomatoid growth in the biopsy
* Other metastasized cancer in the last 5 years
* Patient unable to make an informed decision to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with surgical complications according to Clavien-Dindo grade 2-5 | First year after inclusion
  recorded through chart review at 30 and 90 days after treatment. Complications are summed up in case of retreatment before the 12-month follow-up.
Radiological signs of a residual tumor at the 6-month follow-up | 6-month after inclusion
  Radiological sign of residual tumor at 6-month radiology
Number of postoperative hospitalization days (LOS) | Sum of total after all interventions first year after the first intervention
  Number of postoperative hospitalization days (LOS), i.e., the time the patient has been hospitalized after the procedure until discharge. Hospitalization time is accumulated in case of retreatment within 12 months.

SECONDARY OUTCOMES:
Cancer-specific survival (CSS) | 2, 5 and 10 years after inclusion
  Cancer-specific survival (CSS) is the period from cancer diagnosis to death caused by this cancer diagnosis. CSS will be calculated using Kaplan-Meier estimates and cumulative incidence of cancer-specific death.
Overall survival (OS) | 2, 5 and 10 years after inclusion
  State of survival
Change in eGFR one year after treatment | One year after inclusion
  The study aims to assess kidney function impairment one year after treatment. Blood tests for estimated glomerular filtration rate (eGFR) will be compared with preoperative values to monitor changes. Impaired function is defined as eGFR reduction by ≥20% one year after the procedure compared to measurements before treatment for kidney tumors (10).

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kjellman, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden